CLINICAL TRIAL: NCT06714006
Title: A Phase 1 Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Intravenously Administered PYC-003, a Peptide-phosphorodiamidate Morpholino Oligonucleotide Conjugate, in Healthy Adult Participants and Adult Participants With Confirmed PKD1 Mutation-associated Autosomal Dominant Polycystic Kidney Disease
Brief Title: Phase 1 Study to Evaluate the Safety and Tolerability of Intravenously Administered PYC-003
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: PYC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PYC-003-CL-001
Record Dates: First submitted 2024-11-24; First posted 2024-12-03 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease (ADPKD)
Keywords: PKD1; Autosomal Dominant Polycystic Kidney Disease; ADPKD
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant

STUDY DESIGN:
Intervention Model Description: The study comprises of 2 parts:
  Part A (SAD - Healthy) will be conducted as a randomized, double-blind, placebo-controlled, SAD study to assess the safety, tolerability, PK, PD, and immunogenicity of PYC-003 in healthy adult participants. On Day 1, each participant will receive either PYC-003 or placebo, as a single intravenous infusion.
  Part B (SAD - ADPKD) will be conducted as an open-label SAD study to assess the safety, tolerability, PK, PD, and immunogenicity of PYC-003 in adult participants with confirmed PKD1 mutation-associated ADPKD. On Day 1, each participant will receive PYC-003 as a single IV infusion.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Part A will be randomized, double-blind, placebo-controlled, Single Ascending Dose study.
  Part B will be open-label study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A (SAD - Healthy) (Placebo Comparator): Part A will be conducted as a randomized, double-blend, placebo-controlled, Single Ascending Dose Study to assess the safety, tolerability, Pharmacokinetic, Pharmacodynamic, and immunogenicity of PYC-003 in healthy adult participants
  Interventions: Drug: PYC-003
- Part B (SAD - ADPKD) (Active Comparator): Part B will be conducted as an open-label Single Ascending Dose study to assess the safety, tolerability, Pharmacokinetic, Pharmacodynamic, and immunogenicity of PYC-003 in adult participants with confirmed PKD1 mutation-associated ADPKD.
  Interventions: Drug: PYC-003

INTERVENTIONS:
Drug: PYC-003 — A peptide-phosphorodiamidate morpholino oligonucleotide conjugate administered as a single intravenous infusion

SUMMARY:
This is a Phase 1, First-in-Human study to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD) and immunogenicity of PYC-003 in healthy adult participants and adult participants with confirmed PKD1 mutation-associated Autosomal Dominant Polycystic Kidney Disease (ADPKD) There are 2 parts in this study, i.e. Part A and Part B.

DETAILED DESCRIPTION:
Part A (SAD - Healthy) will be conducted as a randomized, double-blind, placebo-controlled, SAD study to assess the safety, tolerability, PK, PD, and immunogenicity of PYC-003 in healthy adult participants.

The anticipated number of participants across 3 Part A (SAD - Healthy) cohorts is approximately 24 participants.

On Day 1, each participant will receive the investigational product (IP; ie, PYC-003 or placebo), as a single intravenous (IV) infusion. All Part A (SAD - Healthy) cohorts will first dose 2 sentinel participants in a blinded manner on Day 1.

Part B (SAD - ADPKD) will be conducted as an open-label SAD study to assess the safety, tolerability, PK, PD, and immunogenicity of PYC-003 in adult participants with confirmed PKD1mutation-associated ADPKD. The anticipated number of participants across 3 Part B (SAD - ADPKD) cohorts is approximately 18 participants. On Day 1, each participant will receive PYC-003 as a single IV infusion.

ELIGIBILITY:
Key Inclusion Criteria

1. Male or female aged 18 to 65 years (inclusive) at the time of informed consent.
2. ADPKD diagnosis as confirmed by the presence of genetic mutations associated with ADPKD, including, but not limited to, the presence of PKD1 mutation. Note: Where genotyping is not included the medical history for a participant, genotyping may be completed at Pre-Screening.
3. Class 1C, 1D, or 1E per Mayo Imaging Classification System for Predicting Kidney Outcomes in ADPKD (Irazabal et al. 2015) (based upon prior magnetic resonance imaging [MRI] or computed tomography [CT] scan obtained > 6 months prior to Screening, or MRI obtained during Pre-Screening).
4. BMI ≥ 18.0 and ≤ 32.0 kg/m2 and weight ≥ 50 kg.
5. Non-smoker and must not have used any tobacco or nicotine products within 2 months prior to Screening.
6. Estimated glomerular filtration rate (eGFR) ≥ 30 mL/min/1.73 m2 via the CKD EPI 2021 calculation (Inker et al. 2021).

8. Hematology and serum chemistry results at Screening that meet the following criteria:

1. Platelets > 150 × 10^9/L
2. Total white blood cell count > 3.0 × 10^9/L
3. Absolute neutrophil count > 1.5 × 10^9/L
4. Hemoglobin > 110 g/L for females and > 120 g/L for males
5. Total and direct bilirubin < 1.5 × ULN, unless elevated bilirubin is associated with a known benign condition (e.g., Gilbert's syndrome)
6. Alanine aminotransferase (ALT) < 1.5 × ULN
7. Aspartate aminotransferase (AST) < 1.5 × ULN
8. Alkaline phosphatase (ALP) < 1.5 × ULN
9. Gamma-glutamyl transferase < 2 × ULN Note: Screening laboratory testing may be repeated once at the discretion of the PI or designee to confirm out-of-range(exclusionary) results.

Key Exclusion Criteria

1. Presence of potentially confounding genetic mutations (per genotyping by a NATA accredited or equivalent diagnostic laboratory)including, but not limited to, the presence of PKD2, HNF1B, GANAB, IFT140, and/or DNAJB 11 mutations. Note: Where genotyping is not included the medical history for a participant, genotyping may be completed at Pre-Screening.
2. Use of (or anticipated use of) Tolvaptan and/or metformin administration within 30 days prior to the first administration of IP until study completion.
3. Any renal or systemic pathology other than ADPKD or any other condition or prior therapy that in the opinion of the PI or designee would make the participant unsuitable for this study.
4. Has only 1 kidney or has a kidney transplant.
5. History of borderline to low blood magnesium and potassium levels and/or Screening or Day -1 blood magnesium level < 0.7 mmol/L and potassium levels < 3.5 mmol/L.

   Note: Repeat testing (i.e., 1 repeat per parameter) at Screening or Day -1 is permitted for out-of-range values following approval by the PI or designee.
6. Proteinuria > 500 milligrams per 24 hours.
7. Hematuria (urine albumin:creatinine ratio > 30 mg/mmoL, or hematuria > ++ on dipstick, or > 100 cells per high-power field on microscopy)and/or urinary abnormalities at Screening deemed by the PI or designee to be of moderate or higher severity.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
(Part A and B) Number of participants with treatment-related adverse events as assessed by CTCAE V5.0 | 24 weeks
  To evaluate the safety and tolerability of PYC-003 following a single dose administered intravenously to healthy adult participants and adult participants with confirmed PKD1 mutation-associated ADPKD. The incidence, severity, and relatedness of TEAEs and treatment-emergent SAEs will be recorded
(Part A and B) To evaluate the changes in Heart rate via 12-lead ECG (local) following a single dose of PYC-003 administered intravenously | 24 weeks
  To evaluate the safety and tolerability of PYC-003 following a single dose administered intravenously to healthy adult participants and adult participants with confirmed PKD1 mutation-associated ADPKD
(Part A and B) To evaluate the changes in ECG PR interval from baseline via 12-lead ECG (local) following a single dose of PYC-003 administered intravenously | 24 weeks
  To evaluate the safety and tolerability of PYC-003 following a single dose administered intravenously to healthy adult participants and adult participants with confirmed PKD1 mutation-associated ADPKD
(Part A and B) To evaluate the changes in ECG QRS duration from baseline via 12-lead ECG (local) following a single dose of PYC-003 administered intravenously | 24 weeks
  To evaluate the safety and tolerability of PYC-003 following a single dose administered intravenously to healthy adult participants and adult participants with confirmed PKD1 mutation-associated ADPKD
(Part A and B) To evaluate the changes in ECG QT interval from baseline via 12-lead ECG (local) following a single dose of PYC-003 administered intravenously | 24 weeks
  To evaluate the safety and tolerability of PYC-003 following a single dose administered intravenously to healthy adult participants and adult participants with confirmed PKD1 mutation-associated ADPKD
(Part A and B) To evaluate the changes in ECG QTcF interval from baseline via 12-lead ECG (local) following a single dose of PYC-003 administered intravenously | 24 weeks
  To evaluate the safety and tolerability of PYC-003 following a single dose administered intravenously to healthy adult participants and adult participants with confirmed PKD1 mutation-associated ADPKD
(Part A and B) To evaluate the changes in baseline body temperature following a single dose of PYC-003 administered intravenously | 24 weeks
  To evaluate the safety and tolerability of PYC-003 following a single dose administered intravenously to healthy adult participants and adult participants with confirmed PKD1 mutation-associated ADPKD
(Part A and B) To evaluate the changes in baseline systolic and diastolic blood pressure following a single dose of PYC-003 administered intravenously | 24 weeks
  To evaluate the safety and tolerability of PYC-003 following a single dose administered intravenously to healthy adult participants and adult participants with confirmed PKD1 mutation-associated ADPKD
(Part A and B) To evaluate the changes in baseline pulse rate following a single dose of PYC-003 administered intravenously | 24 weeks
  To evaluate the safety and tolerability of PYC-003 following a single dose administered intravenously to healthy adult participants and adult participants with confirmed PKD1 mutation-associated ADPKD
(Part A and B) To evaluate the changes in baseline respiratory rate following a single dose of PYC-003 administered intravenously | 24 weeks
  To evaluate the safety and tolerability of PYC-003 following a single dose administered intravenously to healthy adult participants and adult participants with confirmed PKD1 mutation-associated ADPKD
(Part A and B) To evaluate the changes physically via complete and symptom-directed physical examination following a single dose of PYC-003 administered intravenously | 24 weeks
  To evaluate the safety and tolerability of PYC-003 following a single dose administered intravenously to healthy adult participants and adult participants with confirmed PKD1 mutation-associated ADPKD Complete and symptom-directed physical examinations are to be performed by a licensed physician.
  Complete physical examinations include general appearance, head, ears, eyes, nose, throat, dentition, thyroid, chest (heart, lungs), abdomen, skin, neurological, extremities, back, neck, musculoskeletal, and lymph nodes.
(Part A and B) To evaluate the changes from baseline in serum potassium, serum magnesium, serum sodium, serum osmolality, serum cystatin C, and serum creatinine following a single dose of PYC-003 administered intravenously | 24 weeks
  To evaluate the safety and tolerability of PYC-003 following a single dose administered intravenously to healthy adult participants and adult participants with confirmed PKD1 mutation-associated ADPKD
(Part A and B) To evaluate the changes from baseline in urine potassium, urine magnesium, urine creatinine, and urine osmolality following a single dose of PYC-003 administered intravenously | 24 weeks
  To evaluate the safety and tolerability of PYC-003 following a single dose administered intravenously to healthy adult participants and adult participants with confirmed PKD1 mutation-associated ADPKD
(Part A and B) To evaluate the changes in standard renal and hepatic clinical chemistry parameters following a single dose of PYC-003 administered intravenously | 24 weeks
  To evaluate the safety and tolerability of PYC-003 following a single dose administered intravenously to healthy adult participants and adult participants with confirmed PKD1 mutation-associated ADPKD

SECONDARY OUTCOMES:
(Part A and B) The peak plasma concentration, Cmax of PYC-003 following a single dose administered intravenously | 24 weeks
  This is done to characterize the plasma PK of PYC-003 in participants following a single dose administered intravenously, for both healthy adult participants and adult participants with confirmed PKD1 mutation-associated ADPKD
(Part A and B) The peak plasma concentration, Tmax (time to maximum observed plasma drug concentration) of PYC-003 following a single dose administered intravenously | 24 weeks
  This is done to characterize the plasma PK of PYC-003 in participants following a single dose administered intravenously, for both healthy adult participants and adult participants with confirmed PKD1 mutation-associated ADPKD
(Part A and B) The Plasma PK parameter, t½ (half life) of PYC-003 will be determined following a single dose administered intravenously to adult participants | 24 weeks
  This is done to characterize the plasma PK of PYC-003 in participants following a single dose administered intravenously, for both healthy adult participants and adult participants with confirmed PKD1 mutation-associated ADPKD
(Part A and B) The Plasma PK parameter, AUC0-24 (Area under the plasma concentration versus time curve over the last 24 hour) of PYC-003 will be determined following a single dose administered intravenously | 24 weeks
  This is done to characterize the plasma PK of PYC-003 in participants following a single dose administered intravenously, for both healthy adult participants and adult participants with confirmed PKD1 mutation-associated ADPKD
(Part A and B) Plasma PK parameter, AUC0-inf (extrapolated area under concentration-time curve) of PYC-003 will be determined following a single dose administered intravenously to adult participants | 24 weeks
  This is done to characterize the plasma PK of PYC-003 in participants following a single dose administered intravenously, for both healthy adult participants and adult participants with confirmed PKD1 mutation-associated ADPKD
(Part A and B) The Plasma PK parameter, AUC%extrap (the area under the curve) of PYC-003 will be determined following a single dose administered intravenously | 24 weeks
  This is done to characterize the plasma PK of PYC-003 in participants following a single dose administered intravenously, for both healthy adult participants and adult participants with confirmed PKD1 mutation-associated ADPKD
(Part A and B) The Plasma PK parameter, kel (elimination rate constant) of PYC-003 will be determined following a single dose administered intravenously | 24 weeks
  This is done to characterize the plasma PK of PYC-003 in participants following a single dose administered intravenously, for both healthy adult participants and adult participants with confirmed PKD1 mutation-associated ADPKD
(Part A and B) The Plasma PK parameter, Vz (Volume of distribution) of PYC-003 will be determined following a single dose administered intravenously | 24 weeks
  This is done to characterize the plasma PK of PYC-003 in participants following a single dose administered intravenously, for both healthy adult participants and adult participants with confirmed PKD1 mutation-associated ADPKD
(Part A and B) The Plasma PK parameter, CL (Total drug clearance from plasma) of PYC-003 will be determined following a single dose administered intravenously | 24 weeks
  This is done to characterize the plasma PK of PYC-003 in participants following a single dose administered intravenously, for both healthy adult participants and adult participants with confirmed PKD1 mutation-associated ADPKD

CONTACTS AND LOCATIONS:
Locations (6):
- Australia (6):
  - South Coast Renal, Brockway House, Level 1, Suite 8, 82-86 Queen Street,, Southport, Gold Coast
  - Liverpool Hospital, Clinic G-Reception 133, Level 1, Clinical Building, Burnside Drive, Liverpool, New South Wales
  - Westmead Hospital, Clinical Research Unit, Level 6, B Wing/Building, Hawkesbury Road, Westmead, New South Wales
  - Mater Hospital Brisbane, South Brisbane, Queensland
  - Sunshine Hospital, Western Centre for Health Research and Education, Level 3, 176-190 Furlong Road, Saint Albans, Victoria
  - Linear Clinical Research, Joondalup, Western Australia